CLINICAL TRIAL: NCT06843850
Title: Evaluation of the Effect of Different Irrigation Solutions Used in Regenerative Endodontic Treatment of Necrotic Open Apexed Lower Molar Teeth on Lesion Healing-Randomized Clinical Trial
Brief Title: Lesion Healing After Regenerative Endodontic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ipek Eraslan Akyuz, specialist dentist, TC Erciyes University
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/302
Record Dates: First submitted 2025-01-31; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Apical Periodontitis
Keywords: irrigation solution; lesion healing; regenerative endodontics
MeSH Terms: conditions — Periapical Periodontitis | interventions — Regenerative Endodontics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EDTA (Experimental)
  Interventions: Device: regenerative endodontics
- Citric acid (Experimental)
  Interventions: Device: regenerative endodontics

INTERVENTIONS:
Device: regenerative endodontics — The effect of different irrigation solutions on lesion healing in regenerative endodontics will be compared.

SUMMARY:
Endodontics involves various therapeutic interventions for diagnosing, preventing, and managing pulpal and periradicular pathologies. Root canal treatment, a widely performed procedure, involves removing necrotic pulp tissue and replacing it with a root-filling material, but it limits the tooth's immune defense and regenerative capacity. In immature permanent teeth, pulpal damage can lead to incomplete root formation, increasing the risk of fractures. To address these challenges, regenerative endodontic procedures (REPs) promote tissue regeneration within the root canal using tissue engineering principles.

Despite high success rates, REPs lack a standardized irrigation protocol. Current guidelines recommend using 17% EDTA after low-concentration NaOCl to reduce cytotoxicity and release bioactive molecules. Citric acid has shown promise in in vitro studies as an alternative chelating agent, but direct comparisons with EDTA in clinical settings remain limited. This study aims to bridge this gap by evaluating the long-term effects of EDTA and citric acid on clinical symptoms and lesion healing in REPs.

DETAILED DESCRIPTION:
Endodontics includes various therapeutic interventions to diagnose, prevent, and manage pulpal and periradicular pathologies, including endodontic infections (Duncan et al., 2023). Root canal treatment is a widely performed procedure globally (Leveque et al., 2024) for cases of irreversible pulpitis or pulp necrosis, facilitating the healing of periapical tissues and preventing apical periodontitis. This treatment involves the removal of necrotic pulp tissue and its replacement with a root-filling material. However, despite its effectiveness, conventional root canal therapy is inherently limited in biological activity, as it compromises the tooth's immune defense, vascularization, and regenerative capacity.

Pulpal damage in immature permanent teeth can result from caries, traumatic injuries, or developmental anomalies, leading to pulp necrosis and incomplete root formation (Palma et al., 2017). In such cases, conventional endodontic approaches pose significant challenges due to the high risk of root fractures and extrusion of filling materials, given the presence of thin dentinal walls and open apices (Shah et al., 2008). Furthermore, the lack of adequate root maturation compromises the tooth's structural integrity, increasing its susceptibility to fracture (Bracks et al., 2019). Consequently, novel biomaterials and regenerative strategies have been introduced to address these challenges.

Regenerative endodontic procedures (REPs) have emerged as biologically driven treatments that offer the potential to restore functional dentition by promoting tissue regeneration within the root canal space of immature necrotic teeth (Shamszadeh et al., 2019, Kim et al., 2018). These procedures leverage the principles of tissue engineering, which are fundamental to their long-term efficacy, incorporating key elements such as stem cells, three-dimensional scaffolds, signaling molecules, and a sterile microenvironment (Bracks et al., 2019).

Clinical studies utilizing REPs have yielded promising outcomes, demonstrating high survival and success rates ranging from 95% to 100% (Arslan et al., 2019, Alobaid et al., 2014). Additionally, these studies have reported increased root length, thickness, and apical closure (Shah et al., 2008, Torabinejad and Faras, 2012). Despite these favorable findings, a standardized irrigation regimen for REPs has yet to be established (Shamszadeh et al., 2019). Current clinical guidelines from the American Association of Endodontists (AAo, 2016) recommend the application of 17% ethylenediaminetetraacetic acid (EDTA) following the use of low-concentration sodium hypochlorite (NaOCl).

The inclusion of EDTA is crucial in mitigating NaOCl-induced cytotoxicity while facilitating the liberation of bioactive molecules from dentin (Chae et al., 2018). Moreover, dentin conditioning with EDTA removes the smear layer, thereby exposing growth factors sequestered within the dentin matrix (Bracks et al., 2019). The utilization of chelating agents as a final conditioning step in REP protocols is instrumental in enhancing dentin demineralization, thereby promoting the release of bioactive molecules that can foster the migration, adhesion, and differentiation of stem cells from the periapical region. While EDTA remains the benchmark agent for dentin conditioning in REPs, alternative chelating agents, such as citric acid, have been primarily assessed in vitro and have demonstrated potential to improve cellular responses and growth factor release (Ivica et al., 2019).

A recent systematic review examining both clinical and laboratory-based studies indicated that citric acid enhances smear layer removal and induces a greater release of TGF-β1 compared to other solutions (Gómez-Delgado et al., 2023). However, another systematic review and meta-analysis reported that 10% citric acid resulted in lower TGF-β1 release compared to 10% EDTA (Tavares et al., 2021). However, these prior studies did not directly compare citric acid with EDTA, the standard conditioning agent in REPs, nor were their findings exclusively focused on regenerative endodontic procedures. Consequently, further research is warranted to establish the optimal chelating agent for dentin conditioning in REPs. Since no previous studies have directly compared the effectiveness of EDTA and citric acid in assessing long-term clinical symptoms or their impact on lesion healing, the present study aims to fill this gap and provide more comprehensive evidence on the optimal chelating agent for regenerative endodontic procedures.

ELIGIBILITY:
Inclusion Criteria:

The included patients were healthy (Category: American Society of Anesthesiologists class 1). This study included the necrotic, deeply carious mandibular molars of patients born between 2009 and 2015. Preoperative periapical films of the relevant teeth were evaluated, and teeth determined as Stages 2 and 3 according to the Cvek classification were included in the current study [27].

Exclusion Criteria:

* Patients were excluded if they had a systemic disease or were on systemic corticoste roid therapy, patients reported bruxism or clenching, took analgesics or other drugs that might alter their pain during the last 12 h preoperatively, or had a history of allergic reac tions to any of the medications or materials used. Patients with a tooth with severely curved root canals, vertical root fracture, coronal perforation, calcification or more signifi cant than Grade I mobility, or pocket depth greater than 5 mm were also excluded.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the effects of different irrigation solutions used in regenerative endodontics on lesion healing using surveys | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No